CLINICAL TRIAL: NCT03537794
Title: Characterizing Dopamine D2 and D3 Receptor Binding in Treatment Resistant Depression
Brief Title: Characterizing Dopamine Receptor Binding in Treatment Resistant Depression
Status: Not yet recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Other Study IDs: TPET-01
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment Resistant Depression: Unmedicated Individuals with Treatment Resistant Depression
  Interventions: Diagnostic Test: PET scans
- Major Depressive Disorder: Unmedicated Individuals with Major Depressive Disorder
  Interventions: Diagnostic Test: PET scans
- Healthy Control: healthy controls with no previous psychiatric disorders
  Interventions: Diagnostic Test: PET scans

INTERVENTIONS:
Diagnostic Test: PET scans — PET scans and PHNO scans

SUMMARY:
It is estimated that 30% of individuals with Major Depressive Disorder (MDD) fail to respond to conventional antidepressant medication which accounts for over 1 million Canadians in their lifetime. Treatment resistant depression (TRD) patients also have greater psychiatric and medical comorbidity, poorer quality of life and increased suicidal ideation. Yet, there are few treatment strategies available to target TRD and there is a significant lack of evidence about how TRD differs from treatment-responsive depression. This proposal represents the first study to elucidate the neurobiology of TRD with a focus on dopamine receptor function throughout the brain, in order to inform treatment development and clinical characterization of TRD.The ultimate goal of this unique study is to characterize striatal and extrastriatal dopamine D2 and D3 receptor binding potential in patients with TRD, non-resistant MDD and healthy controls. The primary hypothesis is that TRD patients will exhibit greater D2/D3 receptor binding potential compared to non-TRD patients in the following regions of interest: dorsolateral prefrontal cortex, orbitofrontal cortex, and ventral striatum. Secondarily, non-TRD patients will also demonstrate increased binding potential compared to healthy controls in the same brain regions. Whole brain analyses will allow us to take an exploratory approach to other brain regions that may differentiate TRD from non-TRD patients. Participants will be assessed at St. Michael's Hospital (SMH) and the Centre for Addiction and Mental Health (CAMH), which are within a 10 minute driving distance of each other. There will be 3 study visits following written informed consent. Eligibility will be confirmed at a screening visit at SMH where demographic information, including age, sex, education, and medication history will be obtained, as well as the administration of a structured Mini-International Neuropsychiatric Interview (MINI) for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Axis I diagnoses (Sheehan et al, 2015), and an HRSD-17. Within two weeks of the screening visit, participants will undergo a structural magnetic resonance imaging (MRI) scan at SMH prior to the positron-emission tomography (PET) scan at CAMH. The order of the PHNO scans will be counterbalanced.

ELIGIBILITY:
Inclusion Criteria:

* Key inclusion criteria for the MDD patients:

  * DSM-5 criteria for a Major Depressive Episode (MDE) within a MDD, confirmed through MINI diagnosis (Sheehan et al, 2015)
  * Age between 25 and 55 years
  * Hamilton Depression Rating Scale - 17 item (HRSD-17; Hamilton, 1960) > 14 (moderate to severe symptoms)
  * Free of psychotropic medications for at least 5 half-lives before PET scanning
  * Ability to undergo MRI scanning (absence of metal, pacemakers, etc.)
  * For non-resistant patients: Previous history of response to an antidepressant, in order to increase signal to noise between resistant and non-resistant patients

Key inclusion criteria for the Healthy Controls:

* Ages between 25 and 55 years
* Ability to undergo MRI scanning (absence of metal, pacemakers, etc.)

Exclusion Criteria:

Key exclusion criteria for the MDD patients:

* Pregnancy/lactation
* Medical condition requiring immediate investigation or treatment
* Recent (< 6 months)/current history of drug abuse/dependence
* Lifetime history of psychosis, other Axis I comorbidities are allowable
* Use of any psychotropic use within 5 half-lives before the PET scanning
* For non-resistant patients: Failure of > 2 antidepressant treatments of adequate dose and duration for current MDE.

Key exclusion criteria for the Healthy Controls:

* Pregnancy/lactation
* Medical condition requiring immediate investigation or treatment
* Lifetime history of any psychiatric disorder
* Lifetime history of receiving an antidepressant

Ages: 25 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Participants will be recruited from clinics at St. Michael's Hospital and the Centre for Addiction and Mental Health as well as from research programs at the two sites, which have ongoing MDD clinical trials where patients are required to be unmedicated prior to initiating treatment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dopamine potential | 3 years
  TRD patients exhibit greater D2/D3 receptor binding potential

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: Undecided